CLINICAL TRIAL: NCT01069445
Title: Open Label, Randomized Study of the Impact of Diet on Gut Microbiota, Inflammageing and Oxidative Stress in Elderly People. Potential Benefits of Dietary Advices Alone or Associated to Nutraceutical Food Supplements Argan Oil, VSL#3 Probiotic Blend, 5203-L Fruit Extract Terpene. French Part of a Multicentric European Study
Brief Title: Potential Benefits of Dietary Advices Alone or Associated to Nutraceutical Food Supplements Argan Oil, VSL#3 Probiotic Blend, 5203-L Fruit Extract Terpene
Acronym: RISTOMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2009/08
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Healthy Elderly People
Keywords: diet; probiotics; inflammaging; oxidative stress; gut microbiota; food complements
MeSH Terms: interventions — argan oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diet advices (Active Comparator): will receive the Optimal Diet for Elderly
  Interventions: Behavioral: Optimal Diet
- Diet advices + VSL-3 (Experimental): will receive the Optimal Diet for Elderly + VSL#3® probiotic blend
  Interventions: Dietary Supplement: VSL#3® probiotic blend
- Diet advices + 5203-L (Experimental): will receive the Optimal Diet for Elderly + AISA-5203-L fruit extracted terpene
  Interventions: Dietary Supplement: AISA-5203-L fruit extracted terpene
- Diet advices + Argan oil (Experimental): will receive the Optimal Diet for Elderly + Argan oil
  Interventions: Dietary Supplement: Argan oil

INTERVENTIONS:
Dietary Supplement: VSL#3® probiotic blend — Product should be administrated orally, 2 capsules b.i.d. on an empty stomach (at least 30 min. before lunch and dinner) with a glass of water
  Arms: Diet advices + VSL-3
Dietary Supplement: AISA-5203-L fruit extracted terpene — Product should be administrated orally, the dosage depending from the body weight of the subject enrolled in the study as already stated : 1-2 pills three times a day with a meal and a large glass of water
  Arms: Diet advices + 5203-L
Dietary Supplement: Argan oil — Product should be administrated orally, 25 ml once daily or during the day with a meal (bread, salad …) and a large glass of water
  Arms: Diet advices + Argan oil
Behavioral: Optimal Diet — a dietician will train each subject (or the caregiver) to use the personalized diet on web platform.
  Arms: Diet advices

SUMMARY:
Ageing of the population is a major event in the world. Gerontological/geriatric literature unanimously indicate that physical exercise and diet are at present the two available fundamental approaches to contrast/prevent most of the age associated alterations. In the elderly the inflammageing, the oxidative stress and the alteration of the intestinal microbiota can be influenced by nutritional status and possibly corrected by an appropriate dietetic intervention:

Nowadays the nutraceutical food supplements become an opportunity for the consumer to improve the quality of individual diet for specific needs This study will focus on the development of a specific dietary approach through an E-Health dietary service, associated or not to nutraceutical food supplements intake, to modulate the oxidative stress, inflammageing and gut microflora in the elderly people.

DETAILED DESCRIPTION:
Ageing of the population is a major event in the world. Gerontological/geriatric literature unanimously indicate that physical exercise and diet are at present the two available fundamental approaches to contrast/prevent most of the age associated alterations. In the elderly the inflammageing, the oxidative stress and the alteration of the intestinal microbiota can be influenced by nutritional status and possibly corrected by an appropriate dietetic intervention:

Nowadays the nutraceutical food supplements become an opportunity for the consumer to improve the quality of individual diet for specific needs

ELIGIBILITY:
Inclusion Criteria:

* Age: from 65 to 85 years
* Body Mass Index: 22-30 kg/m2
* ECOG Performance status: WHO performance score 0 to 2
* Absence of known diseases and/or abnormalities of haematological parameters (haematological, inflammatory, metabolic, hepatic and renal diseases)
* The subjects must be able to comply with management of nutraceutical products and with scheduled follow-up
* The subjects must be able to use the computer and to access to the web, by themselves or with the help of a caregiver

Exclusion Criteria:

* History of significant neurologic or psychiatric disorders including dementia, seizures, bipolar disorder
* Geriatric anorexia [less than 2 full meals per day and /or less than one serving of dairy products (milk, cheese, yogurt) per day or two or more servings of legumes or eggs per week or one serving of meat, fish or poultry every day]
* Weight loss > 5% in the last month
* Previous antibiotic treatment within 4 months
* Active infection requiring per OS or IV antibiotics, including active tuberculosis, known and declared HIV, HCV
* Constipation and/or abdominal pain/discomfort that require dietary supplements or medical therapy
* Gastric disease that requires medical therapy (e.g. gastric secretion inhibitory drugs)
* Chronic inflammatory bowel disease (Crohn's disease or ulcerative colitis, diverticulosis, diverticulitis)
* Diabetes mellitus
* Dislipidemia and/or any metabolic disease that requires medical or dietetic treatment
* Myocardial infarction within 6 months prior to study entry, congestive heart disease, uncontrolled cardiac insufficiency, and any current grade 3 or 4 cardio-vascular disorder despite treatment
* Current history of neoplasm except for curatively treated non melanoma skin cancer or in situ carcinoma of the cervix and except for other cancer curatively treated and with no evidence of disease for at least 5 years
* Other sever underlying medical conditions, which could impair the ability of the patient to participate in the study
* Chronic anti-inflammatory therapy with FANS or previous therapy within 20 days from the beginning of the study. The occasional use of anti-inflammatory therapy is not an exclusion criteria, but the use is not allowed within 3 days before the analysis and for more than 8 days/2 months during the study
* Previous (within 15 days) or concomitant treatment that modifies intestinal absorption (e.g. metformine, acarbose in diabetic treatment…)
* Probiotics, prebiotics or simbiotics (yogurt or another functional foods) intake in the last 3 weeks
* Use of food supplements or functional foods such as probiotics, prebiotics, simbiotics, vitamins and minerals different than whose established in this study, is not allowed during the study period or previously within 1 week (except for vitamin D, calcium, vitamin B12)
* Total parenteral nutrition within 4 months
* History of allergy to one of the excipients present in the products under evaluation
* Concomitant or within 4 week period administration of any experimental drug, food supplements or nutraceuticals under investigation
* Subjects clearly intending to withdraw from the study if not randomised in a given arm, or subjects who cannot be regularly followed up for psychological, social, familial or geographic reasons
* Subjects with expected non-compliance to protocol guidelines

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The primary beneficial effect parameter is hsPCR (high-sensitivity C-reactive protein) | 2 months

SECONDARY OUTCOMES:
Inflammageing status: WBC, hemoglobin, ERS, fibrinogen, total cholesterol, triglycerides, insulin, glucose, (and HOMA Index), interleukin-6, TNFα, IL-10, TGF1, IGF-1, adiponectin, lectin, Homocysteine, folic acid and vitamin B12, calprotectin | 2 months
Oxidative stress: plasma total antioxidant capacity by TEAA (Trolox Equivalent Antioxidant Activity), glutathione level, the superoxide dismutase, the glutathione peroxidase, the glutathione reductase and the catalase activities | 2 months
Gut microbiota: expression of 16S ribosomal RNA in bacterial groups from faeces. Ratio between lactobacilli and clostridia bacteria. Real time PCR and PCR DGGE | 2 months
Quality of life: SF-36, GHQ, and daily VAS, ECOG performance status, IADL, Speilbeger Anxiety Scale, CES-D scale | 2 months
Physical performance status (SPPB), muscle function (hand-grip dynamometry), and physical activity level (IPAQ) | 2 months
Compliance to the web diet advices and to the nutraceutical supplement intake (daily VAS) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle BOURDEL-MARCHASSON, Professor, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Pôle de gerontology Clinique Hôpital Xavier Arnozan , University Hospital, Bordeaux, Pessac, France

REFERENCES:
- [Background] Franceschi C, Valensin S, Bonafe M, Paolisso G, Yashin AI, Monti D, De Benedictis G. The network and the remodeling theories of aging: historical background and new perspectives. Exp Gerontol. 2000 Sep;35(6-7):879-96. doi: 10.1016/s0531-5565(00)00172-8. PMID 11053678
- [Background] Wener MH, Daum PR, McQuillan GM. The influence of age, sex, and race on the upper reference limit of serum C-reactive protein concentration. J Rheumatol. 2000 Oct;27(10):2351-9. PMID 11036829
- [Background] Mendall MA, Patel P, Ballam L, Strachan D, Northfield TC. C reactive protein and its relation to cardiovascular risk factors: a population based cross sectional study. BMJ. 1996 Apr 27;312(7038):1061-5. doi: 10.1136/bmj.312.7038.1061. PMID 8616412
- [Background] Devaraj S, O'Keefe G, Jialal I. Defining the proinflammatory phenotype using high sensitive C-reactive protein levels as the biomarker. J Clin Endocrinol Metab. 2005 Aug;90(8):4549-54. doi: 10.1210/jc.2005-0069. Epub 2005 May 17. PMID 15899961
- [Derived] Ostan R, Bene MC, Spazzafumo L, Pinto A, Donini LM, Pryen F, Charrouf Z, Valentini L, Lochs H, Bourdel-Marchasson I, Blanc-Bisson C, Buccolini F, Brigidi P, Franceschi C, d'Alessio PA. Impact of diet and nutraceutical supplementation on inflammation in elderly people. Results from the RISTOMED study, an open-label randomized control trial. Clin Nutr. 2016 Aug;35(4):812-8. doi: 10.1016/j.clnu.2015.06.010. Epub 2015 Jul 15. PMID 26249791
- [Derived] Valentini L, Pinto A, Bourdel-Marchasson I, Ostan R, Brigidi P, Turroni S, Hrelia S, Hrelia P, Bereswill S, Fischer A, Leoncini E, Malaguti M, Blanc-Bisson C, Durrieu J, Spazzafumo L, Buccolini F, Pryen F, Donini LM, Franceschi C, Lochs H. Impact of personalized diet and probiotic supplementation on inflammation, nutritional parameters and intestinal microbiota - The "RISTOMED project": Randomized controlled trial in healthy older people. Clin Nutr. 2015 Aug;34(4):593-602. doi: 10.1016/j.clnu.2014.09.023. Epub 2014 Oct 8. PMID 25453395